CLINICAL TRIAL: NCT06842355
Title: A Multicenter, Phase 2, Dose-Escalation/Dose-Expansion Study of TYRA-300 in Children With Achondroplasia With Open Growth Plates: BEACH301
Brief Title: A Study of TYRA-300 in Children With Achondroplasia: BEACH301
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tyra Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TYR300-201
Record Dates: First submitted 2025-01-29; First posted 2025-02-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TYRA-300 0.125 mg/kg (Experimental): TYRA-300 is provided as sprinkle capsules/mini-tablets. The total dose will be calculated based on the participant's weight. Weight adjustments will be made every 3 months.
  Interventions: Drug: TYRA-300 0.125 mg/kg
- TYRA-300 0.25 mg/kg (Experimental): TYRA-300 is provided as sprinkle capsules/mini-tablets. The total dose will be calculated based on the participant's weight. Weight adjustments will be made every 3 months.
  Interventions: Drug: TYRA-300 0.25 mg/kg
- TYRA-300 0.375 mg/kg (Experimental): TYRA-300 is provided as sprinkle capsules/mini-tablets. The total dose will be calculated based on the participant's weight. Weight adjustments will be made every 3 months.
  Interventions: Drug: TYRA-300 0.375 mg/kg
- TYRA-300 0.50 mg/kg (Experimental): TYRA-300 is provided as sprinkle capsules/mini-tablets. The total dose will be calculated based on the participant's weight. Weight adjustments will be made every 3 months.
  Interventions: Drug: TYRA-300 0.50 mg/kg

INTERVENTIONS:
Drug: TYRA-300 0.125 mg/kg — Initial dose level of TYRA-300 per protocol, subsequent dose level escalations will occur based on criteria outlined in the protocol.
  Arms: TYRA-300 0.125 mg/kg
Drug: TYRA-300 0.25 mg/kg — Subsequent dose level escalations will occur based on criteria outlined in the protocol.
  Arms: TYRA-300 0.25 mg/kg
Drug: TYRA-300 0.375 mg/kg — Subsequent dose level escalations will occur based on criteria outlined in the protocol.
  Arms: TYRA-300 0.375 mg/kg
Drug: TYRA-300 0.50 mg/kg — Subsequent dose level escalations will occur based on criteria outlined in the protocol.
  Arms: TYRA-300 0.50 mg/kg

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and identify potentially effective dose(s) of TYRA-300 in children with achondroplasia with open growth plates.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, open-label, dose-escalation study to determine the safety, tolerability, and identify potentially effective dose(s) of TYRA-300, a fibroblast growth factor receptor (FGFR)-3 selective tyrosine kinase inhibitor, in children 3 to 10 years of age with achondroplasia with open growth plates that will examine three cohorts of children: the Sentinel Safety Cohort, Cohort 1, and Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 to 10 years old (inclusive) at the time of consent.
* Informed consent provided by parent(s) or legal guardian(s). As study participants are less than 18 years old, participants are willing and able to provide written assent (where applicable and required).
* Molecular diagnosis of achondroplasia (FGFR3 G380R).
* Radiographically confirmed open growth plates at Screening, as determined by bone age X-ray.
* Able to stand and ambulate independently.
* Able to take oral medication.
* Sentinel Safety Cohort only: aged 5 to 10 years old (inclusive).
* Cohort 1 only: aged 3 to 10 years old (inclusive) and are naive to prior growth accelerating therapy.
* Cohort 2 only: aged 3 to 10 years old (inclusive) and have received prior growth accelerating therapy.

Exclusion Criteria:

* Presence or history of any concurrent disease or condition that would interfere with study participation, safety evaluations, or any uncontrolled or untreated condition that could impact pediatric growth.
* Diagnosis of endocrine condition that alters calcium/phosphate homeostasis.
* Prior limb lengthening surgery or planned or expected to have limb lengthening surgery while enrolled in the study.
* Taking medications that are strong inhibitors or inducers of cytochrome P450 (Cyp) 3A4.
* History or current evidence of corneal or retinal disorder/keratopathy.
* Presence of guided growth hardware/8 plates. Planned or anticipated orthopedic surgeries.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events as assessed by CTCAE v5.0 | Up to 12 months
Change from baseline in annualized growth velocity (Cohort 1) | 12 months

SECONDARY OUTCOMES:
Change from baseline in annualized growth velocity (Cohort 1) | 6 months
Change from baseline in height z-score (Cohort 1) | 6 and 12 months
Pharmacokinetics: maximum plasma concentration (Cmax) | 15 days
Pharmacokinetics: time to reach maximum plasma concentration (Tmax) | 15 days
Pharmacokinetics: area under the plasma concentration-time curve (AUC) | 15 days
Pharmacokinetics: half-life of TYRA-300 (t1/2) | 15 days
Pharmacokinetics: apparent total clearance (CL/F) | 15 days
Pharmacokinetics: apparent volume of distribution (Vd/F) | 15 days
Change from baseline in annualized growth velocity (Cohort 2) | 6 and 12 months
Change from baseline in height z-score (Cohort 2) | 6 and 12 months
Change from baseline in standing height (cm) | 6 and 12 months
Change from baseline in sitting height (cm) | 6 and 12 months
Change from baseline in upper and lower arm length (cm) | 6 and 12 months
Change from baseline in tibial length (cm) | 6 and 12 months
Change from baseline in femur length (cm) | 6 and 12 months
Change from baseline in arm span proportionality (arm span/height ratio) | 6 and 12 months
Change from baseline in upper segment/lower segment ratio | 6 and 12 months
Change from baseline in elbow extension | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Doug Warner, MD, Study Chair — Tyra Biosciences
Locations (10):
- United States (8):
  - Lundquist Institute for Biomedical Innovation, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Uncommon Cures, Chevy Chase, Maryland
  - University of Missouri, Columbia, Missouri
  - Washington University, St Louis, Missouri
  - Children's Medical Center, Dallas, Dallas, Texas
  - University of Wisconsin-Madison, Madison, Wisconsin
- Royal Children's Hospital, Parkville, Victoria, Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada